CLINICAL TRIAL: NCT00341991
Title: Molecular Epidemiology of Cutaneous Malignant Melanoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902035; 02-C-N035
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Melanoma
Keywords: DNA Repair; Genes; Pigmentation; Skin Cancer; Sun Exposure
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- 1: Cases from hospitals
- 2: Controls from the general populations
- 3: Biological Samples

SUMMARY:
This case-control study was planned to investigate the link of solar radiation with gene damage, host factors, and DNA repair proficiency in cutaneous malignant melanoma (CMM) risk. The hypothesis was that impaired DNA repair proficiency is associated with an increased risk of CMM due to unrepaired DNA damage, particularly in subjects with dysplastic nevi, poor tanning ability or genetic susceptibility.

The study was reviewed as an RO1 Grant from the National Cancer Institute in 1995. Subject enrollment, which included clinical evaluation, epidemiologic questionnaires, and skin and blood sample collection, was completed in 1999 on approximately 180 melanoma cases and 180 controls identified in Italy. The study protocol and consent form both included the measurement of genetic and biochemical factors and DNA repair capacity. DNA repair proficiency was measured in lymphocytes by the host cell reactivation assay, and sun exposure was evaluated by means of a detailed questionaire. Photographs of the back of the subjects were taken to allow nevi count. Minimal erythemal dosage was measured in all subjects to estimate skin sun sensitivity 24 hours after skin's UV-irradiation. Skin color was ascertained on the inner side of the forearm by means of a Minolta chromometer.

The aim of this protocol is to continue analysis of the biological samples already collected, as originally outlined in the study protocol. In particular, we plan to measure polymorphisms in genes that may lead to susceptibility to melanoma. Initially we will concentrate on variation in genes involved in repairing damaged DNA, but plan to look at a broad group of candidate susceptibility genes.

DETAILED DESCRIPTION:
The original case-control study was planned to investigate the link of solar radiation with gene damage, host factors, including also genetic variants, and DNA repair proficiency in cutaneous malignant melanoma (CMM) risk, in subjects from the Mediterranean area, characterized by a wide range of pigmentary characteristics and intense sun exposure. This study was reviewed and funded as an R01 grant from the National Cancer Institute in 1995. Subject enrollment, which included clinical evaluation, epidemiologic questionnaires, and skin and blood sample collection, was completed in 1999 on approximately 180 melanoma cases and 180 controls identified in Italy. The study protocol and consent form both included the measurement of genetic and biochemical factors, and DNA repair capacity. DNA repair proficiency was measured in lymphocytes by the host cell reactiviation assay, and sun exposure was evaluated by means of a detailed questionnaire. Minimal erythemal dosage was measured in all subjects to estimate skin sun sensitivity 24 hours after skin's UVirradiation. Skin color was ascertained on the inner side of the forearm by means of a minolta chromometer.

The aim of this protocol was to continue the analysis of the biological samples and data already collected, as originally outlined in the study protocol. However, the original sample size was small and precluded specific analyses of gene-environment interaction crucial for the understanding of the etiology of melanoma. We have identified other collaborators willing to share their data and sample with us to increase the power for statistical analyses. We obtained approval (amendments to 02-C-N035 approved in November 2006, September 2008, December 2010, and June 2011) to use the DNA samples and data collected in four studies conducted by investigators at the University of L'Aquila, Italy, University of Genoa, Italy, Istituto Valenciano de Oncologia, Valencia, Spain, and the New York University School of Medicine, respectively. We have obtained approval with stipulations in August 2014 to also include samples and data collected from the Papa Giovanni XXII Hospital in Bergamo, Italy and the University of Athens, Greece. We are now responding to the stipulations and asking to further include samples from the University of Padua and the Hospital Clinic of Barcelona within the same study.

We are currently analyzing genes in several pathways, including pigmentation, DNA repair, immune-related functions and those involved in the transition from nevi to melanoma (genes in the cell cycle, telomere, signaling pathways, etc). With the additional samples we plan to conduct a GWAS analysis of melanoma in Mediterranean countries and a molecular analysis of melanoma tissue lesions for an improved classification of the disease and its association with melanoma progression.

ELIGIBILITY:
* Analysis on samples already collected.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases from hospitals; Controls from the general populations
Sampling Method: Non-Probability Sample
Enrollment: 15401 (Actual)
Dates: Start 2001-11-01 (Actual); Primary Completion 2007-09-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Genome-wide association studies, environmental and somatic analyses | Ongoing
  To identify genes, host and environmental factors that lead to susceptibility to melanoma.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Landi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Landi MT, Bauer J, Pfeiffer RM, Elder DE, Hulley B, Minghetti P, Calista D, Kanetsky PA, Pinkel D, Bastian BC. MC1R germline variants confer risk for BRAF-mutant melanoma. Science. 2006 Jul 28;313(5786):521-2. doi: 10.1126/science.1127515. Epub 2006 Jun 29. PMID 16809487
- [Background] Landi MT, Kanetsky PA, Tsang S, Gold B, Munroe D, Rebbeck T, Swoyer J, Ter-Minassian M, Hedayati M, Grossman L, Goldstein AM, Calista D, Pfeiffer RM. MC1R, ASIP, and DNA repair in sporadic and familial melanoma in a Mediterranean population. J Natl Cancer Inst. 2005 Jul 6;97(13):998-1007. doi: 10.1093/jnci/dji176. PMID 15998953
- [Background] Nagore E, Heidenreich B, Rachakonda S, Garcia-Casado Z, Requena C, Soriano V, Frank C, Traves V, Quecedo E, Sanjuan-Gimenez J, Hemminki K, Landi MT, Kumar R. TERT promoter mutations in melanoma survival. Int J Cancer. 2016 Jul 1;139(1):75-84. doi: 10.1002/ijc.30042. Epub 2016 Mar 2. PMID 26875008